CLINICAL TRIAL: NCT00265408
Title: Pilot Study of Aspirin Versus Warfarin for Cervicocephalic Arterial Dissection
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCSD IRB #051253
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2007-03

CONDITIONS: Ischemic Stroke
Keywords: Cervicocephalic Arterial Dissection
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin; Warfarin

ARMS (2):
- aspirin (Experimental)
  Interventions: Drug: aspirin
- warfarin (Experimental)
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: aspirin
  Arms: aspirin
Drug: warfarin
  Arms: warfarin

SUMMARY:
Pilot Study of Aspirin Versus Warfarin for Cervicocephalic Arterial Dissection.

DETAILED DESCRIPTION:
20 patients with cervicocephalic arterial dissection will be randomized to open-label aspirin or warfarin, rate of stroke and adverse events will be endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and imaging diagnosis of cervicocephalic arterial dissection within 3 months.

Exclusion Criteria:

* Any contraindication to aspirin or warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-12; Study Completion 2007-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of stroke by one year. | 1 year

SECONDARY OUTCOMES:
Recurrent dissection by one year. | 1 year
Incidence of TIA by one year. | 1 year
Incidence of major and minor bleeding episodes by one year. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Matt B Jensen, MD, Principal Investigator — UCSD Stroke Center
Locations (1):
- UCSD Medical Center, San Diego, California, United States